CLINICAL TRIAL: NCT02079272
Title: REBECCA Study (RadiothErapy for BrEast Cancer and CArdiotoxicity): Evaluation of Radiation-induced Cardiotoxicity of Adjuvant Radiotherapy With Tomotherapy for Breast Cancer
Brief Title: REBECCA Study (RadiothErapy for BrEast Cancer and CArdiotoxicity)
Acronym: REBECCA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sophie JACOB (Other Government)
Collaborators: Institut de Radioprotection et de Surete Nucleaire (Other Government); Institut Claudius Regaud (Other); University Hospital, Toulouse (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor-Investigator, Sophie JACOB, PhD, Institut de Radioprotection et de Surete Nucleaire
Organization: Institut de Radioprotection et de Surete Nucleaire (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00929-36
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Toxicity Due to Radiotherapy; Breast Cancer; Lesion; Cardiac
Keywords: Tomotherapy; Breast Cancer; Heart; Subclinical cardiac lesions; Myocardial lesions; Coronary lesions; Circulating biomarkers; Ionizing radiation; Heart absorbed doses
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Helical tomotherapy for breast cancer (Other): All women included in REBECCA cohort will be treated with helical tomotherapy for theur breast cancer.
  Their cardiac follow-up will be based on echocardiography, CT coronary angiogram and blood samples
  Interventions: Other: Helical tomotherapy for breast cancer

INTERVENTIONS:
Other: Helical tomotherapy for breast cancer — 1. At baseline, before helical tomotherapy is performed, for each included woman will have:
     * measures of biomarkers of cardiac injury based on blood samples (including CRP, NT-Pro BNP, …, microparticles and miRNA)
     * cardiologic examination including echocardiography for measurement of strain and strain rate
     * a CT coronary angiogram for measurement of coronary plaque indexes
  2. Helical tomotherapy will be performed for all women included in the cohort.
  3. At the end of tomotherapy, follow-up will include:
     * measures of biomarkers: at the end of radiotherapy, 6 months and 24 months after radiotherapy
     * cardiologic examinations including a echocardiography 6 and 24 months after radiotherapy
     * A CT coronary angiogram 24 months after radiotherapy

SUMMARY:
The purpose of this study is to determine whether a new technique of radiotherapy for breast cancer (helical tomotherapy) can induce cardiac toxicity that would be detected in the first two years after treatment. Screening of subclinical cardiac lesions with non-invasive cardiac imaging techniques combined with measures of circulating biomarkers of cardiac tissue lesions and coronary lesions would allow assessing radiation-induced cardiac toxicity at an early stage.

DETAILED DESCRIPTION:
REBECCA study will consist in a monocentric prospective cohort that will include 120 women volunteers treated with adjuvant tomotherapy for breast cancer in the Institut Regaud Claudius-Toulouse (ICR) and followed for 2 years after radiotherapy.

In summary, women aged between 40 and 70 years, surgically treated at ICR for breast cancer and for whom adjuvant radiotherapy with tomotherapy is indicated, with no indication of chemotherapy will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Women treated surgically for left or right breast cancer and for who adjuvant treatment is radiotherapy with irradiation of the breast or chest wall irradiation and possibly lymph node chains,
* Age between 40 and 70 years
* Adjuvant Radiotherapy is helical tomotherapy performed at Institut Claudius Regaud(Toulouse, France)

Exclusion Criteria:

* Indication of adjuvant chemotherapy
* Clinically or radiologically detectable metastasis
* Personal history of coronary artery or myocardial disease
* Personal history of breast cancer or other cancer requiring radiotherapy to the chest
* Contraindications to injection of iodinated contrast ( for CT ) : pregnancy , renal failure, allergy.
* Pregnancy, lactation
* Before radiotherapy, LVEF <50%
* Before radiotherapy, longitudinal strain > - 16 %
* Before radiotherapy,longitudinal strain rate <1% / s
* Before radiotherapy, segmental wall motion abnormality
* Coronary CT before radiotherapy showing that a therapeutic treatment is required

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with subclinical cardiac lesions in myocardial levels and/or coronary levels | within the first 2 years after tomotherapy
  The primary outcome is defined as a decrease of at least 5% in strain or strain rate measures based on cardiac ultrasound exam"2D strain" between the measurement before radiotherapy and measures 24 months after radiotherapy and / or an increase of at least 15% in the average index of coronary plaques measured with CT coronary angiogram between the measurement before radiotherapy and measures 24 months after radiotherapy .

SECONDARY OUTCOMES:
Number of participants with decrease in myocardial contractility (strain or strain rate measured with cardiac ultrasound exam"2D strain") | within the first 6 months after tomotherapy
Number of participants with modified measures of circulating biomarkers | within the first 2 years after tomotherapy (at the end of radiotherapy, 6 months after radiotherapy and 24 months maximum after radiotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Massabeau, MD, Principal Investigator — Institut Claudius Regaud, Toulouse (France); Marie-Odile Bernier, MD, Principal Investigator — Institut de Radioprotection et de Sureté Nucléaire, Fontenay-aux-Roses (France); Jean Ferrières, MD, PhD, Principal Investigator — University Hospital Rangueil, Toulouse (France); Hervé Rousseau, MD, PhD, Principal Investigator — University Hospital Rangueil, Toulouse (France)
Locations (1):
- Institut Claudius Regaud, Toulouse, France